CLINICAL TRIAL: NCT03993808
Title: Improving Cardiovascular Health Through Implementation of a Dietary Approaches to Stop Hypertension (DASH)-Diet-based Multi-component Intervention With Senior Services Programs
Brief Title: DASH Diet Intervention at Senior Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Carter Burden Network (Unknown); Clinical Directors Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RKO-0990
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
Keywords: Nutrition, micro-nutrients, implementation, food insecurity
MeSH Terms: conditions — Hypertension | interventions — Dietary Approaches To Stop Hypertension; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: This is an implementation study, testing whether provision of the evidence-based DASH diet for to community-living seniors as a portion of their daily intake, in the setting of congregate meals at senior centers, coupled with evidence-based home self-blood pressure monitoring, can lead to effective blood pressure lowering.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational/behavioral support for hypertension self efficacy (Experimental): On-site monitoring of pulse, blood pressure, weight, and surveys, at Months 0,1,3,6; Four educational sessions to address: 1) basics about blood pressure (BP); 2) training in home BP monitoring with personal Omron 10 device; 3) information about Dietary Intervention to lower Systemic Blood Pressure (DASH) eating plan, recipes and cooking demonstrations; 4) education about BP medication adherence. Interventions occur on the background of Carter Burden Network's implementation of a DASH-congruent menus for congregant meals for all seniors attending the sites, including those not enrolled in the protocol.
  Interventions: Behavioral: Revision of congregate meal menus and recipes to align with parameters of DASH eating plan; Behavioral: On-site blood pressure monitoring; Behavioral: Home self blood pressure monitoring; Behavioral: Medical adherence education; Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Revision of congregate meal menus and recipes to align with parameters of DASH eating plan — On a programmatic level, congregate meal menus and recipes have been adapted to align with DASH eating. The changes, which include the introduction of additional servings of fruits, vegetables, seeds, grains, replacement of simple or processed carbohydrates with healthier alternatives, introduction of more fish, reduction in added salt, and replacement of animal fats and butter with olive oil, will be phased-in in stages over 6 weeks, concurrent with the start up the study's educational programs addressing nutrition, BP, and medication adherence. The fully DASH-aligned menus will begin by week 7. The dietary intervention affects all seniors eating congregate meals at the center, not only those enrolled in this protocol to study the impact of DASH implementation.
  Other Names: DASH diet
Behavioral: On-site blood pressure monitoring — At baseline (Month 0), and at Months 1, 3, and 6 after the full implementation of the DASH aligned congregate meals, participants will have blood pressure measured by professionals, on-site at the senior center, following established standard procedures. They will receive verbal and written information about their blood pressure results, and encouragement to share the results with their providers.
Behavioral: Home self blood pressure monitoring — Provision of personal Omron 10 home blood pressure monitoring device, training in proper use, and schedule for home self monitoring of BP over the course of the study.
  Other Names: self-measured blood pressure monitoring (SMBP)
Behavioral: Medical adherence education — One required educational session with the community pharmacist to learn about medication adherence strategies
Behavioral: Nutrition Education — One required educational session to review the elements of the DASH eating plan, how to overcome barriers to healthy eating, recipes, cooking demonstrations and materials for household members.

SUMMARY:
The Carter Burden Network (CBN) is an New York City senior services agency, providing vital meal programs for low-income, minority seniors, age 60 and over. In 2016, CBN formed a community-academic partnership with The Rockefeller University (RU) and Clinical Directors Network (CDN) to conduct a Healthy Aging pilot study and found that 84% of participants had high blood pressure, with up to 27% "uncontrolled" using age-adjusted criteria. High blood pressure is a modifiable risk for cardiovascular disease, and has been readily improved in controlled trials by replacement of a typical Western diet with the Dietary Approaches to Stop Hypertension (DASH) diet. The DASH diet has been proven to meaningfully reduce blood pressure in as little as 14 days. However, the DASH diet has not been tested in seniors, in the setting of senior centers. Many seniors attending CBN centers receive close to 40% of their daily nutrition through congregate meals served there. This study tests the effectiveness of implementing the DASH-diet through modification of congregate meals at CBN senior centers to align with DASH, while providing educational and behavioral support, including home self-monitoring of blood pressure, to improve self-efficacy related to blood pressure management. The primary outcome is the change in systolic blood pressure.

DETAILED DESCRIPTION:
The Carter Burden Network (CBN) is an New York City senior services agency, providing vital meal programs for low-income, minority seniors, age 60 and over. Its four senior centers serve 300,000 meals annually through congregate breakfasts and lunches, and home-delivered meals. In 2016, CBN formed a community-academic partnership with The Rockefeller University (RU) and Clinical Directors Network (CDN) to conduct a Healthy Aging pilot study at two of its East Harlem sites, finding that 84% of participants had high blood pressure, with up to 27% "uncontrolled" by age-adjusted criteria. Hypertension continues to be a significant, modifiable, but poorly-controlled contributor to morbidity and mortality from cardiovascular disease (CVD), contributing to stroke, heart attack, renal failure, and cognitive decline, increasing healthcare costs and causing loss of function, independence, and quality of life. Replacement of a typical Western diet with the Dietary Approaches to Stop Hypertension (DASH) diet has been proven to reduce blood pressure in i hypertensive individuals, and individuals with normal blood pressure in as little as 14 days. However, approaches to effective implementation of the DASH diet are untested in community-living seniors.

To address the high cardiovascular risk of uncontrolled hypertension among seniors and introduce innovation into its nutritional program, CBN, RU and CDN designed this two year project to test a DASH-diet-based multi-component intervention to lower blood pressure in two of its senior centers, serving low-income and/or minority seniors. The intervention includes health education, participant input into menu design, redesign of current congregate meals menus to make them with DASH-aligned menus, and home-self monitoring of blood pressure with educational and social support. The primary outcome will be the change in mean systolic blood pressure, measured by health professionals one month after full DASH implementation, compared to baseline. Secondary outcomes include the change in the percentage of seniors with blood pressure in the range of "controlled" by Joint National Committee 8 (JNC-8) guidelines, and the change in blood pressure at three months and at six months.

To optimize acceptance of the changes to menu and recipes, clients will be engaged and provide feedback during the design, implementation and conduct phases of the study. Dietary changes will be planned to incorporate client preferences. Clients will provide feedback weekly on menu acceptability referencing a simple smiley face Likert scale. Educational programs will consist of a series of sessions covering nutritional education including recipes and cooking demonstrations, blood pressure information and training in home self-monitoring with a study-provided blue-tooth enabled Omron 10 device, and information to enhance medication adherence. Participants will have pulse, blood pressure, weight, and behavioral aspects of self-efficacy assessed at baseline, and at Months 1, 3, and 6 of after DASH implementation. Surveys to assess quality of life, food frequency (for compliance with DASH-aligned eating outside of congregate meals), menu satisfaction, medication adherence, and other risks relevant to blood pressure management will be assessed at the same Month 0,1,3,6 time points).

ELIGIBILITY:
Inclusion Criteria:

* A client of the Carter Burden Leonard Covello Senior Center, or the 74th Street Luncheon Club, consuming one or more meals at the center, 4 or more days a week, for at least 3 months, by self report.
* Fluent in English or Spanish
* Currently planning to continue to receive meals at the CBN site (Leonard Covello or Luncheon Club) for the next 6 months

Exclusion Criteria:

* A diagnosis of dementia, early dementia or other cognitive impairment reported by the study participant, the participant's caregiver, CBN staff, or the study team.
* Any condition, that in the opinion of the person obtaining consent, would interfere with the individual's ability to complete the assessments.
* Individuals who rely on a Legal Authorized Representative (LAR)
* Anticipated absence of more than a week, between enrollment and the 1 Month time point

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | One month after implementation of the DASH-aligned congregate meals, compared to Baseline measurement (Month 0) before implementation of dietary or behavioral interventions
  Change in the mean of clients' systolic blood pressure measured at on-site assessments, reported in millimeters of Mercury (mm Hg).
Change in Proportion of individuals with Blood Pressure is in the "controlled" range | One month after implementation of the DASH aligned congregate meals, compared to Baseline measurement (Month 0) before implementation of dietary or behavioral interventions
  The proportion of individuals who blood pressure is within the range "controlled" according to 8th Joint National Committee (JNC-8) guidelines, which for individuals age >60 years, is systolic blood pressure <150 mm Hg, and diastolic blood pressure <90 mm Hg.

SECONDARY OUTCOMES:
Sustainability of Change in Mean Systolic Blood Pressure at 3 months | Month 3 after implementation of DASH meals, compared to Baseline (Month 0), before implementation of any dietary or behavioral changes
  Change in the mean of clients' systolic blood pressure measured at on-site assessments, reported in millimeters of Mercury (mm Hg)
Sustainability of Change in Mean Systolic Blood Pressure at 6 months | Month 6 after full implementation of DASH meals, compared to Baseline (Month 0), before implementation of any dietary or behavioral changes
  Change in the mean of clients' systolic blood pressure measured at on-site assessments, reported in millimeters of Mercury (mmHg)
Enhanced self efficacy - self monitoring | up to Month 1
  Mean frequency of home blood pressure self-monitoring (number of measurements/week)
Cognitive and behavioral change - change in medication adherence self-efficacy | 1 Month after full implementation of dietary changes, compared to Baseline measure
  Change in mean score on Medication Adherence Self-Efficacy Scale (MASES-R) - this survey/scale asks participants how confident they are they can adhere to prescribed medications in 15 different settings that challenge adherence; responses are captured on a 4 point scale from 1-not at all sure, 2-a little sure, 3-fairly sure, and 4-extremely sure. Higher scores are better.
Client acceptance of meals | 1 month after full implementation of dietary changes, compared to Baseline before implementation of any dietary or behavioral changes
  Mean Likert scale score (smiley card) score for DASH-aligned meals; Clients (participants) complete a meal evaluation card once a week, to reflect acceptance of recent menu offerings. The card asks, "Overall, How were the meals this week?" and asks the participant to rate the meals using a 5-point rating scale that ranges from unacceptable meals represented by a deeply frowning red face (1), through intermediates of a mildly frowning orange face (2), neutral expression yellow face (3), slightly smiling light green face (4), to a highly acceptable meal represented by a broadly smiling dark green face (5). Higher scores are better than lower values.
DASH-concordance of meals | During the first month of full implementation of dietary changes, compared to Baseline before implementation of any dietary or behavioral changes
  This measure reflects to what degree the meals as served during the intervention, were DASH-aligned, according to the recommendations of the DASH eating adapted for the designed study menus. This concordance is expressed as the number of the 8 food group requirements satisfied (defined in the DASH eating plan and adapted for the study menus) by the meals as provided. The DASH eating plan identifies 8 groups: 1-Grains, 2-vegetables, 3-fruits, 4-fat-free/low fat milk and milk products, 5-lean meats, poultry and fish, 6-nuts, seeds and legumes, 7-fats and oils, 8-sweets and added sugar. The higher the score, the more DASH-concordant the meal. This outcome will report the mean daily meal DASH-concordance, e.g." 7.5 food group requirements satisfied." For components that allow for weekly requirements rather than daily requirements, (e.g. nuts/seeds) the score for the week (requirement satisfied - yes/no) will be applied to each day within that week.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda G Kost, MD, Principal Investigator — The Rockefeller University
Locations (1):
- Carter Burden Network Leonard Covello Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashemi A, Vasquez K, Guishard D, Naji M, Ronning A, George-Alexander G, Vasquez D, Sylvester C, Pagano W, Khalida C, Coffran C, Ezeonu T, Fofana K, Bielopolski D, Vaughan R, Qureshi A, Tobin JN, Kost RG. Implementing DASH-aligned Congregate Meals and Self-Measured Blood Pressure in two senior centers: An open label study. Nutr Metab Cardiovasc Dis. 2022 Aug;32(8):1998-2009. doi: 10.1016/j.numecd.2022.05.018. Epub 2022 May 31. PMID 35752539